CLINICAL TRIAL: NCT04148885
Title: One-arm, Multi-center Clinical Trial of Paclitaxel (Albumin-binding) Combined With Carboplatin for Castration-resistant Prostate Cancer
Brief Title: A Trial of Paclitaxel (Albumin-binding) for Castration-resistant Prostate Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Qi Li, Executive director of cancer center, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSPC-KAL-PC-01
Record Dates: First submitted 2019-10-29; First posted 2019-11-04 (Actual); Last update posted 2019-11-04 (Actual); Status verified 2019-10

CONDITIONS: Castration-resistant Prostate Cancer
Keywords: castration-resistant prostate cancer; paclitaxel (albumin-binding); carboplatin
MeSH Terms: interventions — 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- nab-paclitaxel + Carboplatin (Experimental): nab-paclitaxel at 260 mg/m^2 on days 1; Carboplatin AUG=5, d1, 21 days in one cycle, 3 cycles in total
  Interventions: Drug: nab-paclitaxel; Drug: carboplatin

INTERVENTIONS:
Drug: nab-paclitaxel — Patients firstly receive nab-paclitaxel 100 mg/m^2 (iv, 30 minutes) on days 1, 8, and 15 for 3 weeks, followed by one week without treatment. Treatment repeats every 4 weeks for up to 6 circles in the absence of disease recurrence or unacceptable toxicity.
  Other Names: Abraxane
Drug: carboplatin — Patients secondly receive carboplatin AUC=5 (iv, 30 minutes) on days 1 for 3 weeks, followed by one week without treatment. Treatment repeats every 4 weeks for up to 6 circles in the absence of disease recurrence or unacceptable toxicity.
  Other Names: Paraplatin; Carboplat; Ercar

SUMMARY:
One-arm, multi-center clinical trial of paclitaxel (albumin-binding) combined with carboplatin for castration-resistant prostate cancer

DETAILED DESCRIPTION:
Prostate cancer is one of the most common malignant tumors of the male genitourinary system. In 2017, the American Oncology Society will report that 161,360 new prostate cancers were estimated, accounting for 21% of male tumors, ranking first in male new tumors; 26,730 death, cancer death. The rate is second only to bronchial lung cancer and colorectal cancer. In China, although the incidence of prostate cancer is lower than the world epidemiological level, the incidence of prostate cancer in China has shown an increasing trend in recent years. The latest statistics from the National Cancer Center 2017, the incidence of male prostate cancer is 2.4%, which is a male malignant tumor. Seventh place in the disease. The taxane drug docetaxel showed good anti-tumor activity in castration resistant prostate cancer (CRPC) patients, and paclitaxel combined with carboplatin also had a certain effect on CRPC. However, in clinical practice, patients with prostate cancer are mostly old, often accompanied by other underlying diseases, poor physical status, and poor tolerance in the use of docetaxel and paclitaxel. Albumin-bound paclitaxel has more tumor-targeted enrichment than traditional paclitaxel and is less toxic. Therefore, this study intends to explore the efficacy and safety of albumin-bound paclitaxel combined with carboplatin in the treatment of CRPC, providing a reference for the treatment options of CRPC in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years, Male;
* diagnosed as prostate cancer by histopathology or cytology;
* Confirmed as castration-resistant prostate cancer: 1 interval 1 week, 3 consecutive PSA minimum values increased by >50%; 2 serum testosterones <50ng/dl or <1.7nmol/L [Guide of the Chinese Urological Association (2015) The diagnostic criteria of CRPC];
* There are no other concurrent anti-cancer treatments (including local radiotherapy, systemic chemotherapy, and molecular targeted therapy) or previous treatment history;
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2;
* The estimated survival period is more than 3 months;
* having at least one measurable lesion according to the RECIST 1.1 tumor evaluation criteria;
* No obvious signs of hematological disease, ANC≥1.5×109/L, platelet count≥100×109/L, Hb≥90g/L, WBC≥3.0×109/L, and no bleeding tendency before enrollment;
* Liver function test: total bilirubin (TBIL) ≤1.5 times the upper limit of normal value, alanine aminotransferase (ALT), aspartate aminotransferase (AST) are ≤2.5 times the upper limit of normal value, if due to liver metastasis, the above indicators ≤5 times the upper limit of normal value; renal function test: serum creatinine (Cr) ≤ 1.5mg/dl, or calculated creatinine clearance rate ≥50ml/min;
* Understand the circumstances of this study, patients and/or legal representatives voluntarily agree to participate in the trial and sign informed consent.

Exclusion Criteria:

* • Have a birth plan during the clinical trial;

  * Patients with brain metastases;
  * Severe cardiovascular diseases such as cerebrovascular accidents occurring within 6 months, myocardial infarction, hypertension that cannot be controlled after drug intervention, unstable angina pectoris, heart failure (NYHA 2-4), and arrhythmia requiring drugs Intervention;
  * Dementia, mental state changes or any mental illness that may interfere with understanding or making informed consent or completing a questionnaire;
  * Subjects with ≥1 peripheral neuropathy according to CTCAE V version 4.03;
  * Allergy or hypersensitivity history of the drug or drug ingredient used in this test;
  * Excluding other malignant tumors, cured basal cell carcinoma of the skin or squamous cell carcinoma of the skin or any other part of the carcinoma in situ;
  * Have received any other test drug treatment or participated in another interventional clinical trial within 30 days of the screening period;
  * The investigator believes that it is not suitable for inclusion.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2019-11 (Estimated); Primary Completion 2020-07 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Prostate specific antigen (PSA) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months
  PSA was effective: PSA decreased by ≥ 50% for more than 4 weeks, and there was no evidence of clinical and imaging progression; PSA progression: PSA increased more than 25% of baseline or baseline during chemotherapy, and the absolute value was ≥ 5 ng/ml.

SECONDARY OUTCOMES:
ORR | From date of enrollment (after curative resection) until the date of death from any cause, assessed one month during therapy and 3 months thereafter
  Objective Response Rate
TTF | From date of enrollment (after curative resection) until the date of death from any cause, assessed one month during therapy and 3 months thereafter
  Time to treatment failure
OS | From date of enrollment (after curative resection) until the date of death from any cause, assessed one month during therapy and 3 months thereafter
  Overall survival